CLINICAL TRIAL: NCT04993547
Title: Peers' and Parent's Presence During Collective Nasopharyngeal COVID-19 Testing Amongst Pupils: A Cluster-Randomized Controlled Trial
Brief Title: Cluster-RCT Collective Nasopharyngeal COVID-19 Testing Amongst Pupils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BAD/DV/2021/BC-09709; BUN6702021000301 (Other: Ghent University Hospital)
Record Dates: First submitted 2021-08-04; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-03

CONDITIONS: Peer Group; Parents
Keywords: Public Health; Pediatric; Nasopharyngeal; Collective testing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parents present, peers present (Experimental): The children are accompanied by their parents during the COVID-19 testing, and a visible covid-19 swab test waiting line is set-up enabling the children to observe their peers being tested.
  Interventions: Other: Parent and peer presence
- Parent present, peers absent (Active Comparator): The children are also accompanied by their parents, but a covered COVID-19 swab test waiting line is set-up whereby the children are unable to observe their peers being tested.
  Interventions: Other: Parent and peer presence
- Parents absent, peers present (Active Comparator): Parents are absent during the COVID-19 testing, and a visible COVID-19 swab test waiting line is set-up enabling the children to observe their peers being tested.
  Interventions: Other: Parent and peer presence
- Parents absent, peers absent (Active Comparator): Parents are absent, and a covered COVID-19 swab test waiting line is set-up whereby the children are not able to observe their peers being tested.
  Interventions: Other: Parent and peer presence

INTERVENTIONS:
Other: Parent and peer presence — Does the presence of fellow pupils and parents improves a pupil's resistance to undergo a nasopharyngeaal swab test?

SUMMARY:
Does the presence of fellow pupils and parents improves a pupil's resistance to undergo a nasopharyngeaal swab test?

DETAILED DESCRIPTION:
In order to control the outbreak of cluster infections on school during the COVID-19 pandemic, regular rounds of collective nasopharyngeal swab testing were organized. However, it is unclear under which circumstances nasopharyngeal swab testing is better accepted by young children. Due to the closing of schools, and the different logistic situations in schools, a natural pragmatic RCT formed. In some cases, children could observe their peers before having their own test, while for others the view was blocked. Also, sometimes parents would be present during a test procedure when the school was closed, while they were not present when the school was open. To date, it is unclear whether these two variable elements influence a child's resistance to be tested. Therefore a cluster-randomized controlled trial with testing site as the unit of randomisation will be set-up. Four conditions will be tested. On the individual level, the resistance of their peers before their own testing will be taken into account. The aim of the study is to compare whether (1) the visibility of nasopharyngeal swab testing on their peers and (2) the presence of their parents impacts a child's resistance towards the test. Additionally, the impact of whether or not their peers resisted the test impact predicts the likelihood of their own resisting behaviour.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a nasopharyngeal COVID-19 swab test

Exclusion Criteria:

-

Ages: 30 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 952 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
test resistance | 1 day
  resistance for swab testing

CONTACTS AND LOCATIONS:
Overall Officials: Simon Malfait, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No